CLINICAL TRIAL: NCT00611741
Title: The Role of Cortical Glutamate and GABA in Brains Osmotic Regulation: A Pilot Study in Healthy Volunteers and in Patients With Schizophrenia
Brief Title: The Effect of Plasma Osmolality on Brain Glutamate
Acronym: MRS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Handan Gunduz-Bruce, Assistant Clinical Professor, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 0612002149
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2012-08

CONDITIONS: Schizophrenia
Keywords: MRS, glutamate, osmolality
MeSH Terms: conditions — Schizophrenia | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug intervention, longitudinal (Experimental): Furosemide and Na supplements
  Interventions: Drug: furosemide, Na supplements

INTERVENTIONS:
Drug: furosemide, Na supplements — furosemide 20 mg, Na supplements 8g in divided doses/day for 5 days

SUMMARY:
This study is designed to test the hypothesis that plasma osmolality is linked with cortical glutamate concentrations in the brain. It also investigates whether the glutamate response in schizophrenia is enhanced compared to healthy controls.

ELIGIBILITY:
Inclusion criteria for healthy controls

1. Ages of 21-45 years from all ethnic backgrounds.
2. Male or female.
3. Written informed consent.
4. Female subjects will be studied during the follicular phase of their menstrual cycle.*

Exclusion criteria for healthy controls

1. DSM-IV diagnosis of psychotic, anxiety, mood disorder.
2. A history of significant medical/neurological disease. Unstable medical condition based on EKG, vital signs, physical examination and laboratory work-up (CBC with differential, SMA-7, LFTs, TFTs, UA, Utox, Urine pregnancy test, folic acid, B12 levels).
3. History of allergies to drugs such as sulfa, multiple adverse drug reactions or known allergy to furosemide.
4. Any medication that in the opinion of the PI could interfere with either the safety of the study and/or the outcome measures, such as over the counter cough suppressants or antihistamines.
5. History of major psychiatric disorder in first-degree relatives.
6. Current substance abuse/dependency determined by plasma and urine toxicology.
7. Current treatment with medications with psychotropic effects.
8. Current pregnancy, unsatisfactory birth control method report for females.
9. Education < 12th grade.
10. Non-English speaking.

Inclusion criteria for patients with schizophrenia

1. Ages of 21-45 years from all ethnic backgrounds.
2. Male or female.
3. Written informed consent.
4. DSM-IV diagnosis of schizophrenia or schizoaffective disorder.
5. For treated patients: The patient has been on a stable dose of medications (antipsychotics, antidepressants) for the past month and does not require a change of medications or dose adjustment at study entry.
6. For untreated patients: Has refused to be treated with medications, maintains regular clinic appointments with the clinicians, and does not pose an imminent danger to himself or others.
7. Female subjects will be studied during the follicular phase of their menstrual cycle*.

Exclusion criteria for patients with schizophrenia

1. A history of significant medical/neurological disease. Unstable medical condition based on EKG, vital signs, physical examination and laboratory work-up (CBC with differential, SMA-7, LFTs, TFTs, UA, Utox, Urine pregnancy test, folic acid, B12 levels).
2. Orthostatic systolic blood pressure change>20 mmHg or orthostatic pulse change>20 bpm.
3. History of polydipsia/hyponatremia**.
4. History of allergies to drugs such as sulfa, multiple adverse drug reactions or known allergy to furosemide.
5. Any medication that in the opinion of the PI could interfere with either the safety of the study and/or the outcome measures, such as over the counter cough suppressants or antihistamines.
6. Current use of lithium (lithium directly interferes with electrolyte balance).
7. Currently on clozapine as clozapine may interfere with brain water regulation (Leadbetter and Shutty, 1994).
8. Current substance abuse/dependency determined by plasma and urine toxicology.
9. Current treatment with benzodiazepines or mood stabilizers (these medications can alter glutamate transmission).
10. Current pregnancy, unsatisfactory birth control method report for females.
11. IQ < 70 as determined by Wechsler Abbreviated Scale of Intelligence.
12. Non-English speaking

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-03; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Cortical glutamate concentration | Baseline and endpoint

SECONDARY OUTCOMES:
Cognitive function | Baseline and end point

CONTACTS AND LOCATIONS:
Overall Officials: Handan Gunduz-Bruce, M.D., Principal Investigator — Yale University
Locations (1):
- 34 Park Street, CMHC, New Haven, Connecticut, United States